CLINICAL TRIAL: NCT06719583
Title: Black and African Americans Connections to Parkinson's Disease (BLAAC PD) a Project of the Global Parkinson's Genetics Program (GP2)
Brief Title: Black and African Americans Connections to Parkinson's Disease (BLAAC PD)
Acronym: BLAAC PD
Status: Recruiting | Type: Observational
Sponsor: Michael J. Fox Foundation for Parkinson's Research (Other)
Collaborators: National Institutes of Health (NIH) (NIH); University of Chicago (Other); University of Alabama at Birmingham (Other); Rush University (Other); Washington University School of Medicine (Other); Medical University of South Carolina (Other); University Hospitals Cleveland Medical Center (Other); Louisiana State University Health Sciences Center Shreveport (Other); University of Florida (Other); University of Maryland (Other); The University of Texas Health Science Center, Houston (Other); Ochsner Health System (Other)
Responsible Party: Sponsor
Other Study IDs: BLAAC PD
Record Dates: First submitted 2024-12-02; First posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Parkinson Disease
Keywords: genetics; racial health disparities
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood or saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Participants with Parkinson's Disease: Data collected from these participants include demographic information and family health history. Participants may also complete a physical exam. Participants also complete a smell test and contribute a blood or saliva sample for genetic analyses.
- Control Participants: Data collected from these participants include demographic information and family health history. Participants also complete a smell test and contribute a blood or saliva sample for genetic analyses.

SUMMARY:
BLAAC PD is a research study to understand what Parkinson's disease looks like for Black and African American communities.

BLAAC PD is happening at research centers around the United States. The study is part of the Global Parkinson's Genetics Program (GP2). GP2 is a research project working to transform understanding of the genetics of Parkinson's disease and make that knowledge globally relevant.

DETAILED DESCRIPTION:
Research studies have found connections between genes and Parkinson's disease (PD). But those results have mostly come from studies with non-Black or African American volunteers. BLAAC PD aims to learn more about gene changes that may cause Parkinson's in Black and African American people. Study volunteers at sites across the United States will attend one visit and will give either a blood or saliva sample, complete a smell test, and may be asked to complete a physical exam. This new data could lead to future Parkinson's tests and treatments for Black and African American people and it may help better understand disease in other groups, too.

This pioneering initiative will fill a gap of knowledge about PD in Black and African American people.

ELIGIBILITY:
Inclusion Criteria for Control Participants:

* Ability to provide informed consent
* Age 18 years or older
* Self-identify as Black or African American

Exclusion Criteria for Control Participants:

* Diagnosis of Parkinson's Disease and/or neurological condition
* Familial history of PD and/or neurodegenerative or psychiatric conditions
* Unknown family history of PD and/or neurodegenerative or psychiatric conditions
* Any conditions that, in the investigator's opinion, preclude the individual's ability to carry out study activities
* If submitting a saliva sample, nothing by mouth (food, drink, gum, tobacco, or smoking) for 30 minutes prior to sample collection

Inclusion Criteria for Participants with a Diagnosis of PD:

* Ability to provide informed consent
* Age 18 years or older
* Self-identify as Black or African American
* Meet the Movement Disorder Society's clinical diagnostic criteria for Parkinson's disease

Exclusion Criteria for Participants with a Diagnosis of PD:

- If submitting a saliva sample, nothing by mouth (food, drink, gum, tobacco, or smoking) for 30 minutes prior to sample collection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Black Americans and African Americans with Parkinson's Disease or without a history of Parkinson's (control volunteers).
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2020-11-16 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Explore novel risk factors and characterization | 5 years
  To explore novel risk factors and characterization of known genetic risk factors contributing to Parkinson's disease risk in the Black and African American population.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Singleton, PhD, Principal Investigator — National Institutes of Health (NIH)
Locations (12):
- United States (12):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Florida, Gainesville, Florida
  - Rush University, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Louisiana State University Health Sciences Center Shreveport, Shreveport, Louisiana
  - University of Maryland, Baltimore, Maryland
  - Kaiser Permanente Midatlantic States, Rockville, Maryland
  - Washington University in St. Louis, St Louis, Missouri
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Texas Health Science Center, Houston, Houston, Texas